CLINICAL TRIAL: NCT03017911
Title: Prospective Observational Study on Picclines' Complications at Brest Hospital
Brief Title: COMPLI-PICC: Study on Picclines' Complications
Acronym: COMPLI-PICC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: COMPLI-PICC
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: PICC Line Placement
Keywords: PICC Line; Complications; Thrombosis; Infection
MeSH Terms: conditions — Thrombosis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PICC Lines: All patients included in this study have undergone PICC Line placement before enrollment.
  Interventions: Procedure: Piccline

INTERVENTIONS:
Procedure: Piccline

SUMMARY:
This is a prospective monocentric study of PICC Line complications use in 5 medical and one surgical units of Brest Medical University Hospital.

To evaluate the incidence of the following complications: infections, thromboses, mechanical and hemorrhagic, at month 3 post-intervention.

Also evaluating:

* the management of these PICC Line related complications,
* risk factors for such complications,
* and the mortality-related outcomes.

DETAILED DESCRIPTION:
All eligible patients fulfilling the inclusion criteria, after PICC Line placement, will receive oral and written patient information describing the study deployment and follow-up. Patients will be followed up until PICC Line removal if it occurs during the first 3 months after placement or until death if it occurs during the first 3 months, or during 3 months in the absence of complications.

* Infectious complications are described in accordance with IDSA 2009 guidelines and include bloodstream infection, endocarditis, local infection and septic thrombophlebitis.
* Thrombotic complications are defined as symptomatic, deep, or superficial venous thrombosis, confirmed by Ultrasound and Echo-Doppler or asymptomatic venous thrombosis diagnosed fortuitously.
* Mechanical complications are defined as impairments related to PICC Line device: occlusion, rupture, accidental removal.
* Hemorrhagic complications are defined as hematoma or bleedings of puncture site.

In the event of PICC Line-related complications, patient will be followed up for an additional 3 months, from the date of complication diagnosis, i.e. maximum follow-up duration of 6 months.

Each week during the first month, then once monthly during the follow-up (i.e. W1, W2, W3, W4, M2, M3, +/- M4, M5, M6), all patients data related to the PICC Line retention or removal, use and all its related complications will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 yo
* Patients > 18 yo hospitalized in internal medicine, pneumology, nutrition, oncology, hematology, and cardiac and vascular surgery - who underwent PICC Line placement between October 10, 2016 and March 9, 2017

Exclusion Criteria:

* Patients hospitalized in other units than those cited above
* Patients verbal refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 yo from internal medicine, pneumology, nutrition, oncology, hematology, and cardiac and vascular surgery - who underwent PICC Line placement between October 10, 2016 and March 9, 2017 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Complication in patient with piccline | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Safdar N, Maki DG. Risk of catheter-related bloodstream infection with peripherally inserted central venous catheters used in hospitalized patients. Chest. 2005 Aug;128(2):489-95. doi: 10.1378/chest.128.2.489. PMID 16100130
- [Background] Chopra V, Ratz D, Kuhn L, Lopus T, Chenoweth C, Krein S. PICC-associated bloodstream infections: prevalence, patterns, and predictors. Am J Med. 2014 Apr;127(4):319-28. doi: 10.1016/j.amjmed.2014.01.001. Epub 2014 Jan 17. PMID 24440542
- [Background] Chemaly RF, de Parres JB, Rehm SJ, Adal KA, Lisgaris MV, Katz-Scott DS, Curtas S, Gordon SM, Steiger E, Olin J, Longworth DL. Venous thrombosis associated with peripherally inserted central catheters: a retrospective analysis of the Cleveland Clinic experience. Clin Infect Dis. 2002 May 1;34(9):1179-83. doi: 10.1086/339808. Epub 2002 Apr 3. PMID 11941543
- [Background] Vidal V, Muller C, Jacquier A, Giorgi R, Le Corroller T, Gaubert J, Champsaur P, Bartoli J, Moulin G. [Prospective evaluation of PICC line related complications]. J Radiol. 2008 Apr;89(4):495-8. doi: 10.1016/s0221-0363(08)71453-7. French. PMID 18477956